CLINICAL TRIAL: NCT05415618
Title: Clinical and Ultrasonographic Evaluation of Manual Lymphatic Drainage and Nerve Mobilization Techniques in Patients Diagnosed With Mild-Moderate Carpal Tunnel Syndrome
Brief Title: Ultrasonographic Evaluation of the Effectiveness of Different Techniques
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-14/01
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Ultrasound Evaluation of the Effect of Manual Lymph Drainage; Effect of Manual Lymph Drainage on Carpal Tunnel Syndrome
Keywords: ultrasonographic evaluation; carpal tunnel syndrome; manual lymph drainage; edema; pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Edema; Pain | interventions — Manual Lymphatic Drainage; Splints

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kontrol group (Active Comparator)
  Interventions: Device: splint
- MLD group (Experimental)
  Interventions: Other: Manual lymphatic drainage
- Nerve gliding group (Experimental)
  Interventions: Other: Nerve gliding

INTERVENTIONS:
Other: Manual lymphatic drainage — Manual lymphatic drainage will be applied 5 days a week for about 15 minutes every day for 4 weeks.
  Arms: MLD group
Device: splint — In splint treatment, a volar-supported splint that keeps the wrist in a neutral position will be preferred and it will be recommended to both groups to be used only at night for 4 weeks.
  Arms: Kontrol group
Other: Nerve gliding — Median nerve gliding exercises as a home exercise program will be performed by the patient 5 days a week for 4 weeks. It will be performed in 6 different consecutive positions of the hand and wrist.
  Arms: Nerve gliding group

SUMMARY:
Carpal tunnel syndrome (CTS) occurs as a result of compression of the median nerve under the transverse ligament along the carpal tunnel. The main cause of median nerve compression and carpal tunnel syndrome is increased volume in the carpal tunnel. The pressure that edema puts on the nerve must be controlled in the early period. Edema that persists beyond the inflammatory process can contribute to the fibrotic stage, delay healing, and even cause complications such as pain and stiffness. Manual lymphatic drainage (MLD) is a specialized technique that involves gentle massage techniques and follows lymphatic pathways from proximal to distal and then from distal to proximal. On the basis of this concept; Increasing circulation by stimulating the lymph system, removing biochemical residues, reducing edema and pain, and regulating sympathetic and parasympathetic system responses. It is known that MLD rapidly regulates lymphatic circulation by creating a change in interstitial fluid pressure, thus preventing even arthrofibrotic tissue that may form after a traumatic situation, reducing edema that predisposes to pain, and increasing mobility. Nerve gliding exercises are another method used in treatment. By providing a sliding movement of the tendons and median nerve in the distal-proximal direction, mobilization of the surrounding soft tissues is achieved and dynamic ischemia is terminated. The aim of this study is to determine the effectiveness of manual lymphatic drainage and nerve mobilization on clinical and ultrasonographic findings in carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate carpal tunnel syndrome on electrodiagnostic examination
* Being between 20-55 years old
* Volunteering to participate in the treatment to be given

Exclusion Criteria:

* Have a systemic inflammatory disease
* Having any disease that may cause polyneuropathy, such as diabetes mellitus
* Cognitive impairment
* Receiving psychotherapy
* Having a pacemaker
* illiterate
* Having a disease affecting the central nervous system
* Having a hearing problem
* Any skin disease that would contraindicate manual lymphatic drainage
* Arterial or venous circulatory disorders that would contraindicate manual lymphatic drainage
* NSAID drug use

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-04-12 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic Evaluation | 20 minutes
  Median nerve diameter measurements and depths of the participants will be made by USG with a multifrequency (7-15 MHz) linear probe. With USG, the median CBF and its depth will be measured distally from the level of the scaphoid bone (wrist; carpal tunnel level) and the midpoint of the forearm.
Evaluation of symptom severity and functional status | 10 minutes
  It will be assessed with the Boston Carpal Tunnel Questionnaire (BCTQ). 1. The symptom severity scale (BCTQSS) has 11 items that evaluate pain, paresthesia, and weakness. 2. The functional status scale (BCTQ-FS) evaluates the ability to perform manual activities with 8 items. Each item evaluates the increasing severity of symptoms or difficulty with a higher score.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Science University Hospital, Kütahya, Turkey (Türkiye)